CLINICAL TRIAL: NCT05432180
Title: Human Milk Nutrients and Infants' Health Outcomes in South China
Status: Completed | Type: Observational
Sponsor: Huilian Zhu (Other)
Responsible Party: Sponsor-Investigator, Huilian Zhu, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: MUAI-2022
Record Dates: First submitted 2022-06-20; First posted 2022-06-27 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Faeces were retented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to investigate the associations between human milk nutrients and infants' health outcomes in China.

DETAILED DESCRIPTION:
Human milk components are beneficial to the growth and development of infants, such as phospholipids, gangliosides, sialic acids, choline, oligosaccharide and so on. However, studies on the associations between human milk components and infants' outcomes are limited. Therefore, this study is designed to investigate the relationship between Chinese human milk components and the growth and development of infants.

ELIGIBILITY:
Inclusion Criteria:

* age 4-5 years
* healthy children
* breastfeeding between 0 to 400 days of age
* human milk components in human milk being determined
* sign informed consent

Exclusion Criteria:

* children with severe chronic diseases, such as tumor, severe digestive diseases, kidney diseases
* gestational diabetes, hypertension and other metabolic diseases
* children with mental system diseases
* children with congenital and genetic diseases
* children with infectious diseases, eg, upper respiratory tract infection or diarrhea
* antibiotic or other drugs influencing intestinal flora being taken within 45 days
* Withdraw withdraw informed consent serious violation of the scheme no longer meet the research criteria because of health factors or accidents

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children of this study will be recruited from lactating women provided human milk samples before.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
The growth of children | 18 month
  The physical growth and body composition of children will be checked by physical examination.
The cognitive development of children | 18 month
  The brain developments of children will be obtained by the Griffith Developmental Assessment Scale.
Gut microbiota | 6 month
  Gut microbiota of children will be examined by the analysis of 16S rDNA and metagenomic.

SECONDARY OUTCOMES:
General demographic materials | 14 month
  The general demographic materials of parents and children will be obtained by questionnaire.
Dietary and lifestyle information | 3 month
  Dietary and lifestyle information of children will be obtained by questionnaire.
Behavior problems | 18 month
  The behavior problems are collected by Child Behavior Checklist.
Allergic assessment | 18 month
  Allergic assessments of children will be conducted by questionnaire.
Sleep assessment | 18 month
  Sleep assessment of infants will be conducted by The Children's Sleep Health Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Huilian Zhu, Professor, Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang MT, Lan QY, Pan C, Huang SY, Huang ZH, Li MC, Li Z, Li F, Li X, Zou JP, Chen HQ, Qiu YZ, Song S, Mao YY, Zhu HL. Long-term cognitive benefits of human milk phospholipids in breastfed children at preschool age: results from MUAI study. Eur J Nutr. 2025 Sep 23;64(7):283. doi: 10.1007/s00394-025-03801-y. PMID 40986082